CLINICAL TRIAL: NCT02744027
Title: Dynamic Contrast Enhanced MR Lymphangiogram Imaging of Lymphatic Anomalies (LA)
Brief Title: Imaging of Lymphatic Anomalies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-012331
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Gorham Disease; Lymphatic Diseases; Lymphangiomatosis
Keywords: Generalized Lymphatic Anomaly; Kaposiform Lymphangiomatosis; Dynamic Contrast Enhanced Magnetic Resonance Lymphangiogram; Magnetic Resonance Imaging
MeSH Terms: conditions — Osteolysis, Essential; Lymphatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dynamic Contrast Enhanced Magnetic Contrast Imaging (Other): Dynamic Contrast Enhanced Magnetic Resonance (MR) Lymphangiogram and heavy T2 Magnetic Resonance imaging data will be evaluated for abnormal lymphatic perfusion of the lung parenchyma. Abdominal and thoracic lymphatic malformations will be characterized by location, number, size, relationship to other organs and perfusion patterns in order to create a basis of imaging classification of lymphatic abnormalities (LA). Subjects will undergo both Dynamic Contrast Enhanced Magnetic Resonance Lymphangiogram (DCMRL) and Heavy Weighted T2 Imaging.
  Interventions: Other: Dynamic Contrast Enhanced Magnetic Resonance Lymphangiography (DCMRL); Other: Heavy Weighted T2 Imaging (T2W); Other: Lymph Node Access

INTERVENTIONS:
Other: Dynamic Contrast Enhanced Magnetic Resonance Lymphangiography (DCMRL) — Following completion of the T2 lymphatic mapping, contrast agent administered will be calculated based on weight. Investigators will use dosage of 0.1cc/kg of contrast which will be injected by hand simultaneously into each lymphatic node (LN) at a rate of 0.5-1 cc per min. One minute after the injection, scanning will be initiated using high spatial and temporal resolution magnetic resonance angiography (syngo time-resolved angiography with stochastic trajectories [TWIST]) sequence. The sequence parameters will be adjusted with a time delay such that a complete volume will be acquired approximately every 20-60 seconds. This will be followed by additional scans with a high-resolution navigator gated 3-dimensional flash inversion recovery (IR) sequence. In all subjects the scan area covered the neck, chest, and abdomen as caudal as feasible.
Other: Heavy Weighted T2 Imaging (T2W) — Magnetic Resonance imaging (MRI) will be performed and T2W MRI lymphatic mapping will be performed using a respiratory navigated and cardiac gated 3 dimensional turbo spin echo sequence with pre-set parameters. Scan time varies from 2-5 min depending upon the size of the subject.
Other: Lymph Node Access — The procedure will be performed under sedation and anesthesia if participants are aged 16 or under. The procedure will be performed with local anesthesia for participants aged over 16 years old.
  Using ultrasound guidance two inguinal lymph nodes (one each side) will be directly accessed with 25-gauge spinal needles attached to a short connector tubing. A shallow angle for puncture will be used to create a long subcutaneous tract to assist in stabilizing the needle. A small amount of an oil-based contrast or water soluble contrast will be injected under fluoroscopy guidance to confirm the correct position of the needles inside the lymph nodes. After stabilizing the needle, the subjects will be transferred into the MRI suite.

SUMMARY:
Lymphatic Anomalies (LA) is characterized by proliferation of lymphatic tissue causing deterioration of pulmonary function. Understanding changes in lymphatic anatomy in these patients is hindered by the difficulty of imaging the lymphatic system. Dynamic Contrast Enhanced MR Lymphangiogram (DCMRL) may be useful in investigating pathological changes in the lymphatic system.

DETAILED DESCRIPTION:
Lymphatic anomalies (LA) are a spectrum of rare diseases classified into lymphatic tumors and malformations. Complicated LA cases in the past have been called lymphangiomatosis because of varied disseminated involvement including soft tissue and viscera such as the spleen, liver and bone. Pleural effusions and pericardial effusions are often associated with these lesions. These are now classified into different phenotypes such as Generalized Lymphatic Anomaly (GLA), Gorham's Stout Disease (GSD) and Kaposiform Lymphangiomatosis (KLA). These complicated phenotypes can cause massive osteolysis causing a morbidity and mortality from infection or paralysis or worsening pulmonary function and effusions (GSD, GLA, KLA).

The major cause of mortality and morbidity in these patients is the deterioration of pulmonary function by chronic chylous effusions and progressive interstitial lung disease. Unfortunately, little is known about biomarkers, risk stratification or the pathophysiology of this progression. The understanding of changes in patients' lymphatic anatomy with LA is hindered by the difficulty of imaging the lymphatic system. Dynamic Contrast Enhanced MR Lymphangiogram (DCMRL) is a technique that has recently been developed, allowing dynamic MR imaging of the lymphatic system by injecting gadolinium contrast agent in the groin lymph nodes.

This technique has been previously used to identify pathological lymphatic perfusion of the lung parenchyma in patients with plastic bronchitis and neonatal chylothorax. Based on these imaging findings, a treatment algorithm has been designed and used to successfully treat the majority of those patients with these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with Lymphatic Anomalies (GLA, KL, Gorham disease) with radiological and or pathological confirmation of lung involvement will be considered for the study.
* Girls > 11 y.o. with a negative urine pregnancy test and contraception use.
* Registration in the International Lymphangiomatosis and Gorham's Disease Alliance (LGDA) Patient Registry or referral by a physician.

Exclusion Criteria:

* Subjects with contraindications to contrast enhanced MRI: allergy to gadolinium imaging agents, impaired renal function (GFR<30) and presence of paramagnetic objects.
* Claustrophobia or contraindications to sedation/anesthesia
* Uncorrectable coagulopathy (bleeding disorders).
* Pregnant or lactating females.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Describe lymphatic anatomy of participants with lymphatic anomalies (LA) | 2 Days
  The primary endpoint will be the description of lymphatic anatomy assessing if participants have a single or branched Thoracic Duct.

SECONDARY OUTCOMES:
Development of a classification system for lymphatic flow | 2 days
  Development of a classification system based on retrograde or anterograde flow of lymphatic fluid.
Description of Lymphatic malformations in participants with lymphatic anomalies | 2 days
  Assessing if lymphatic malformation are present or absent in participants with lymphatic anomalies.

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Dori, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Itkin M, Rabinowitz DA, Nadolski G, Stafler P, Mascarenhas L, Adams D. Abnormal Pulmonary Lymphatic Flow in Patients With Lymphatic Anomalies and Respiratory Compromise. Chest. 2020 Aug;158(2):681-691. doi: 10.1016/j.chest.2020.02.058. Epub 2020 Mar 24. PMID 32220591